CLINICAL TRIAL: NCT04868513
Title: Enhancing Effect of the Application of 1% Chlorhexidine Varnish With Silane Fluoride and Oral Health Promotion on the Streptococcus Mutans Counts Reduction in Pregnant Women and on Early Mother-infant Transmission
Brief Title: Streptococcus Mutans Reduction Early Mother-infant Transmission
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biochemical and Microbiology Laboratory, Faculty of Dentistry, Autonomous University of San Luis Pot (Other)
Responsible Party: Principal Investigator, Marine Ortiz Magdaleno, Research professor, Biochemical and Microbiology Laboratory, Faculty of Dentistry, Autonomous University of San Luis Pot
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Oral health promotion
Record Dates: First submitted 2021-04-14; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pregnant Women
Keywords: chlorhexidine varnish; silane fluoride; Streptococcus mutans; vertical transmission
MeSH Terms: interventions — Fluor Protector; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Random clinical trial of parallel groups
Who Masked: Investigator
Masking Description: Two groups were formed assigning 28 women to each intervention group. G-I received 0.1% silane fluoride applied as varnish in each visit. G-II women's teeth were coated with 0.1% silane fluoride and 1% chlorhexidine. For the primary culture, CRT Bacteria® system (Ivoclar-Vivadent™) was used for the growth and identification of cariogenic Streptococci.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Pregnant women to whom applied silane fluoride (Experimental): We applied 0.1% silane fluoride (Fluor Protector, Ivoclar Vivadent AG™) as varnish in all teeth on all faces as a promotion strategy on the reduction of S. mutans.
  Interventions: Drug: Pregnant women to whom applied silane fluoride
- Pregnant women to whom applied silane fluoride + 1% chlorhexidine (Experimental): We applied 0.1% silane fluoride (Fluor Protector, Ivoclar Vivadent AG™) and 1% chlorhexidine (Cervitec, Ivoclar Vivadent AG™), both applied as varnish, with a 1 min interval between applications, in all teeth on all faces, using the standardized technique indicated by the manufacturer as a promotion strategy on the reduction of S. mutans.
  Interventions: Drug: Pregnant women to whom applied silane fluoride + 1% chlorhexidine
- Children of the pregnant women to whom it was applied silane fluoride (No Intervention): The children not given any intervention, they were only subjected to a microbiological and clinical examination.
- Children of the pregnant women to whom it was applied silane fluoride + 1% chlorhexidine (No Intervention): The children not given any intervention, they were only subjected to a microbiological and clinical examination.

INTERVENTIONS:
Drug: Pregnant women to whom applied silane fluoride — Pregnant women who received 0.1% silane fluoride applied as varnish in the teeth.
  Other Names: Fluor Protector, Ivoclar Vivadent AG™
  Arms: Pregnant women to whom applied silane fluoride
Drug: Pregnant women to whom applied silane fluoride + 1% chlorhexidine — Pregnant women who received silane fluoride + 1% chlorhexidine applied as varnish in the teeth.
  Other Names: Fluor Protector, Ivoclar Vivadent AG™ + 1% chlorhexidine
  Arms: Pregnant women to whom applied silane fluoride + 1% chlorhexidine

SUMMARY:
Evidence exists on the vertical transmission of Streptococcus mutans from the mother to her children. This transmission can be prevented by maintaining maternal oral health during pregnancy.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the enhancing effect of 1% chlorhexidine varnish together with silane fluoride re-mineralizing varnish and oral health promotion strategy on the reduction of S. mutans counts in saliva of pregnant women and the early mother-infant transmission until the first six months of age of the newborn. Methods: An open, random clinical trial of parallel groups was performed. 56 pregnant women free of caries were studied prospectively and longitudinally since the third trimester of gestation until 6 months after giving birth, the newborns were also assessed until reaching 6 months of age. Two groups were formed assigning 28 women to each intervention group. G-I received 0.1% silane fluoride applied as varnish in each visit. G-II women's teeth were coated with 0.1% silane fluoride and 1% chlorhexidine. For the primary culture, CRT Bacteria® system (Ivoclar-Vivadent™) was used for the growth and identification of cariogenic Streptococci. Identification of S. mutans was performed through PCR. The DNA of the isolates identified molecularly as S. mutans was used for a second PCR reaction using the arbitrary primer OPA-O2 to determine the homology among the samples of isolated bacteria from the mother-child pair.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester with a normal and healthy pregnancy.
* Ages ranged from 18 to 45 years
* Free of caries (if caries were present, they were treated before enrolling them in the study).

Exclusion Criteria:

-Non-pregnant women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In pregnant women
Enrollment: 58 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Caries prevalence assessment in pregnant womens | Basal measurement, at the beginning of the third trimester of gestation.
  For this purpose, the Decayed, Missing, and Filled Teeth Index was used to measure the prevalence of caries. This index is based on in-field clinical examination of individuals by using a probe, mirror and cotton rolls, and simply counts the number of decayed, missing (due to caries only) and restored teeth the number of participants with prevalence of caries will be reported.
Streptococcus mutans levels identified in pregnant womens | Basal measurement, at the beginning of the third trimester of gestation.
  In this measurement was identified the S. mutans counts in the saliva of pregnant women after the applications of 1% chlorhexidine varnish together with the application of silane fluoride re-mineralizing varnish or only with the application of silane fluoride, was reported the distribution of cariogenic Streptococcus levels in mothers.
Streptococcus mutans levels identified in pregnant womens | Three months after the birth of the child.
  In this measurement was identified the S. mutans counts in the saliva of pregnant women after the applications of 1% chlorhexidine varnish together with the application of silane fluoride re-mineralizing varnish or only with the application of silane fluoride, was reported the distribution of cariogenic Streptococcus levels in mothers.
Streptococcus mutans levels identified in pregnant womens | Six months after the birth of the child
  In this measurement was identify the S. mutans counts in the saliva of pregnant women after the applications of 1% chlorhexidine varnish together with the application of silane fluoride re-mineralizing varnish or only with the application of silane fluoride. Will be reported the distribution of cariogenic Streptococcus levels in mothers.
Genotypes of the isolates of S. mutans in pregnant womens. | Three months after the birth of the child.
  The genotypes describes an organism's complete set of genes, in this study, was determined the homology among the samples of isolated bacteria from the mother-child pair. The molecular PCR test was implemented for the identification. Will be reported the % of S. mutans genotypes isolated from the mothers of both groups to the strains isolated from the newborns.
Streptococcus mutans levels identified in childrens | Three months after the birth of the child.
  In this measurement was identified the S. mutans counts in the saliva of the children. Will be reported the distribution of cariogenic Streptococcus levels in the children.
Streptococcus mutans levels identified in children | Six months after the birth of the child.
  In this measurement was identified the S. mutans counts in the saliva of the children. Will be reported the distribution of cariogenic Streptococcus levels in the children.
Genotypes of the isolates of S. mutans in children. | Three months after the birth of the child.
  The genotypes describes an organism's complete set of genes, in this study was determined the homology among the samples of isolated bacteria from the mother-child pair, was reported the % of S. mutans genotypes isolated from the children.

IPD SHARING:
Plan to Share IPD: No